CLINICAL TRIAL: NCT00854854
Title: Evaluating the Safety and Efficacy of Combination Therapy With FOLFOX-4 and TKcell Therapy Versus FOLFOX-4 Alone in Patients With Recurrent, Unresectable and Advanced Gastric Cancer
Brief Title: Efficacy Study of TKcell in Advanced Gastric Cancer
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Binex (Industry)
Responsible Party: Park, Eun-Jin / RN, CRM(clinical research manager)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BX-TK-001
Record Dates: First submitted 2009-02-27; First posted 2009-03-03 (Estimated); Last update posted 2009-05-18 (Estimated); Status verified 2009-03

CONDITIONS: Advanced Gastric Cancer
Keywords: NKCell; FOLFOX-4; gastric cancer
MeSH Terms: conditions — Stomach Neoplasms | interventions — Folfox protocol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Control (No Intervention): * Oxaliplatin infusion (100mg/m2) on days 1 and 15 (every 2 weeks)
  * 5-FU bolus + infusions (400 mg/m2) on days 1, 2, 15 and 16
  * LV infusions (200 mg/m2) on days 1, 2, 15 and 16
- Active (Active Comparator): Infusion of TKCell(autologous activated lymphocyte) over 2x10^9 cells, IV route, 7 times
  and chemotherapy schedule
  Interventions: Biological: TKCell

INTERVENTIONS:
Biological: TKCell — TKCell 150ml IV for 7times after each FOLFOX-4 regimen :
  From the second cycle of FOLFOX4(start Day1),TKCell is administered in Day3 and Day8.In the third cycle of FOLFOX4(Day1),TKCell is administered in Day3 and Day8.In the fourth cycle of FOLFOX4(Day1),TKCell is administered in Day8.In the fifth cycle of FOLFOX4(Day1),TKCell is administered in Day8.In the sixth cycle of FOLFOX4(Day1),TKCell is administered in Day8
  Other Names: NKCell; FOLFOX-4
  Arms: Active

SUMMARY:
The purpose of this study is to determine efficacy of NKCell combined FOLFOX-4 chemotherapy in gastric cancer

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent.
* Diagnosis of histologically confirmed adenocarcinoma of the gastric
* ECOG performance status of 0 - 2
* At least one definite measurable lesion(s): ≥ 1 cm on spiral CT scan or ≥2cm in physical examination
* Adequate liver, renal, bone marrow functions as evidence by the following; Absolute neutrophil count > 1.5 x 109/L; platelets > 7.5 x 109/L; Bilirubin less than 2 mg/dL ASAT and/or ALAT < 5 UNL; serum creatinine ≤ 2 ULN
* Minimum life expectancy of 12 weeks
* Effective contraception for both male and female subjects if the risk of conception exists

Exclusion Criteria:

* Brain metastasis and/or leptomeningeal disease (known or suspected)
* Previous chemotherapy for gastric cancer except adjuvant treatment with progression of disease documented > 6 months after end of adjuvant treatment.
* Previous oxaliplatin-based chemotherapy
* Surgery (excluding diagnostic biopsy) or irradiation within 4 weeks prior to randomization and chemotherapy
* HIV antibody (+), Chronic hepatitis
* Uncontrolled infection
* Concurrent or previous chronic systemic immune therapy, targeted therapy, hormonal therapy not indicated in the study protocol except for contraception
* Clinically relevant coronary artery disease, history of myocardial infarction, high risk of uncontrolled arrhythmia
* Known hypersensitivity reaction to any of the components of the treatment.
* Pregnancy (absence to be confirmed by ß-hCG test) or lactation period
* Participation in another clinical study within the 30 days before randomization
* Significant disease which, in the investigator's opinion, would exclude the subject from the study

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 94 (Actual)
Dates: Start 2009-01; Primary Completion 2010-01 (Estimated); Study Completion 2010-07 (Estimated)

PRIMARY OUTCOMES:
Determine response rate | within study period

SECONDARY OUTCOMES:
Determine safety of combination,time to treatment failure, overall survival time | within study period

CONTACTS AND LOCATIONS:
Overall Officials: Seok-Goo Cho, M.D, Ph.D, Principal Investigator — The Catholic Medical Center
Locations (1):
- The catholic University of korea, Banpo-dong, Seoul, South Korea

REFERENCES:
- See also: Click here for more information about this study. — http://www.bi-nex.com/